CLINICAL TRIAL: NCT01833221
Title: Study of the Reinnervation of Facial Muscles After Lengthening Temporalis Myoplasty
Brief Title: Reinnervation of Facial Muscles After Lengthening Temporalis Myoplasty
Acronym: FacialReinn
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study reach enough significance at the intermediary analysis
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-159
Record Dates: First submitted 2013-04-12; First posted 2013-04-16 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2014-04

CONDITIONS: Facial Paresis
Keywords: facial palsy; lengthening temporalis myoplasty; neurotization of facial muscles
MeSH Terms: conditions — Facial Paralysis | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neurotized facial muscle patients (Experimental): injection of 1% lidocaine, 2mL for facial nerve block
  Interventions: Drug: injection of 1% lidocaine, 2mL for facial nerve block

INTERVENTIONS:
Drug: injection of 1% lidocaine, 2mL for facial nerve block — injection with a fine needle of 2mL lidocaine in close contact of the facial nerve trunk
  Other Names: facial nerve block following the O'Brien modified technique

SUMMARY:
The purpose of this study is to determine the physiology of nerve healing and the neurotization of the facial muscles after lengthening temporalis myoplasty.

DETAILED DESCRIPTION:
The investigators want to study the physiology of nerve healing after lengthening temporalis myoplasty done for facial nerve impairment. The investigators already observed few cases of spontaneous neurotization and the investigators want to check the nerve command of the facial muscles. Clinical and photographic evaluations will be performed before and after a facial nerve block using 1% lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* patient who were operated for a facial paralysis by the lengthening temporalis myoplasty procedure in the University Hospital of Caen and who present signs of contraction of the facial muscles on the plasy side after the procedure.

Exclusion Criteria:

* Patient with contraindications to the injection of lidocaine
* Patient treated with beta-blocker
* Patient on anti-coagulants
* Pathology cause of facial paralysis evolving
* Pregnant or lactating
* Patient incapacitated adult
* Patient undergoing another study at the same time

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Facial muscle contraction after nerve block | 30 minutes after lidocaine injection
  clinical and photographical study will be performed before and after neve block and relative contractibility state will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Labbé, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- Centre Hospitalier Universitaire, Caen, Basse-normandie, France

REFERENCES:
- [Background] Cheney ML, McKenna MJ, Megerian CA, West C, Elahi MM. Trigeminal neo-neurotization of the paralyzed face. Ann Otol Rhinol Laryngol. 1997 Sep;106(9):733-8. doi: 10.1177/000348949710600903. PMID 9302902
- [Background] Fournier HD, Denis F, Papon X, Hentati N, Mercier P. An anatomical study of the motor distribution of the mandibular nerve for a masseteric-facial anastomosis to restore facial function. Surg Radiol Anat. 1997;19(4):241-4. doi: 10.1007/BF01627866. PMID 9381330
- [Background] Godwin Y, Tomat L, Manktelow R. The use of local anesthetic motor block to demonstrate the potential outcome of depressor labii inferioris resection in patients with facial paralysis. Plast Reconstr Surg. 2005 Sep 15;116(4):957-61. doi: 10.1097/01.prs.0000178043.15510.75. PMID 16163078
- [Background] Guerreschi P, Labbe D, Carluer L, Drillet C, Benateau H. [Manktelow's test for the use of botulic toxin]. Ann Chir Plast Esthet. 2008 Feb;53(1):59-62. doi: 10.1016/j.anplas.2007.04.010. Epub 2007 Jun 27. French. PMID 17600609
- [Background] Labbe D, Huault M. Lengthening temporalis myoplasty and lip reanimation. Plast Reconstr Surg. 2000 Apr;105(4):1289-97; discussion 1298. PMID 10744217
- [Background] Lifchez SD, Matloub HS, Gosain AK. Cortical adaptation to restoration of smiling after free muscle transfer innervated by the nerve to the masseter. Plast Reconstr Surg. 2005 May;115(6):1472-9; discussion 1480-2. doi: 10.1097/01.prs.0000160266.81504.71. PMID 15861049
- [Background] Petropoulos AE, Cheney ML. Induction of facial muscle neurotization by temporalis muscle transposition: literature review and animal model evaluation using horseradish peroxidase uptake. J Otolaryngol. 2000 Feb;29(1):40-6. PMID 10709171
- [Background] Schimek F, Fahle M. Techniques of facial nerve block. Br J Ophthalmol. 1995 Feb;79(2):166-73. doi: 10.1136/bjo.79.2.166. PMID 7696239